CLINICAL TRIAL: NCT05498233
Title: Open Randomized Cross-over Two-period Study on Comparative Pharmacokinetics and Bioequivalence of Doxylamine + Pyridoxine, Enteric-soluble Film-coated Tablets, 10 mg + 10 mg (Valenta Farm, Russia) in Healthy Volunteers in Fasted Conditions
Brief Title: Pharmacokinetics and Bioequivalence of Doxylamine + Pyridoxine, Film-coated, Enteric-soluble Tablets, and Diclectin, Delayed Release Tablets, in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DIP-05-01-2022
Record Dates: First submitted 2022-08-09; First posted 2022-08-12 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Pregnancy Related; Nausea
MeSH Terms: conditions — Nausea | interventions — dicyclomine, doxylamine, pyridoxine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RT-sequence (Other): Group 1 (14 volunteers, RT sequence) will take 2 tablets of Diclectin in Period 1 and 2 tablets of Doxylamine + Pyridoxine in Period 2
  Interventions: Drug: Doxylamine + Pyridoxine
- TR-sequence (Other): Group 2 (14 volunteers, sequence TR) will take 2 tablets of Doxylamine + Pyridoxine in Period 1 and 2 tablets of Diclectin in Period 2.
  Interventions: Drug: Doxylamine + Pyridoxine

INTERVENTIONS:
Drug: Doxylamine + Pyridoxine — A single dose of R or T drug in each of 2 periods of the study in fasted conditions

SUMMARY:
The study aimed for:

1. Comparative assessment of pharmacokinetic parameters and bioequivalence of the drug Doxylamine + Pyridoxine, enteric-soluble film-coated tablets, 10 mg + 10 mg (Valenta Pharm JSC, Russia), and Diclectin, delayed-release tablets, 10 mg + 10 mg (registrant: Tzamal Bio-Pharma, Israel, manufacturer: Duchesnay Inc, Canada), in healthy volunteers in fasted conditions.
2. Comparative evaluation of the safety of the drug Doxylamine + Pyridoxine, enteric-soluble film-coated tablets, 10 mg + 10 mg (Valenta Pharm JSK, Russia), and Diclectin, delayed-release tablets, 10 mg + 10 mg (registrant: Tzamal Bio-Pharma, Israel, manufacturer: Duchesnay Inc, Canada), based on the analysis of adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary and handwritten informed consent form signed by a healthy volunteer to participate in the study before any of the study procedures.
2. Women of reproductive age (18 to 49 years inclusive, according to World Health Organization criteria).
3. Verified diagnosis "healthy" (absence of abnormalities according to clinical, laboratory, instrumental methods of examination stipulated by the protocol).
4. Blood pressure (BP) level: systolic blood pressure (SBP) from 100 to 139 mmHg, diastolic blood pressure (DBP) from 60 to 89 mmHg (inclusive).
5. Heart rate (HR) from 60 to 90 bpm (inclusive).
6. Respiratory rate (HR) from 12 to 18 bpm (inclusive).
7. Body temperature of 36 to 36.9°C (inclusive).
8. Body mass index (BMI) is 18.5 ≤ BMI ≤ 30 kg/m2, and the body weight must be ≥ 45 kg.
9. Consent to use adequate methods of contraception throughout the study and for 30 days after completion, negative pregnancy test.
10. Volunteers must behave adequately, coherent speech must be observed.

Exclusion Criteria:

1. A history of allergic reactions.
2. Drug intolerance of active and/or excipients included in the study drugs in the anamnesis.
3. Chronic diseases of the cardiovascular, lymphatic, respiratory, nervous, endocrine, digestive, musculoskeletal, covering, immune systems, as well as of the urogenital system and hematopoietic organs.
4. Values of standard laboratory and instrumental indices beyond the limits of local laboratory norms.
5. History of gastrointestinal surgery (except appendectomy at least 1 year before screening).
6. Diseases/conditions that the investigator believes may affect the absorption, distribution, metabolism, or excretion of the study medication.
7. Acute infectious disease less than 4 weeks prior to screening.
8. Taking drugs that have a significant effect on hemodynamics and drugs that affect liver function (barbiturates, benzodiazepines, omeprazole, cimetidine, etc.) for less than one month before screening.
9. Regular intake of drugs less than 2 weeks before screening and one-time intake of drugs less than 7 days before screening.
10. Donating blood or plasma less than 3 months before the screening visit.
11. Use of hormonal contraceptives less than 2 months before the screening visit.
12. Using depot injections of any medications less than 3 months prior to the screening visit.
13. Pregnancy or lactation, positive pregnancy test.
14. Participation in another clinical trial less than 3 months before screening or concurrently with this study.
15. Taking more than 10 units of alcohol (1 unit of alcohol is equivalent to 330 ml of beer, 150 ml of wine, or 40 ml of spirits) in the week in the last month before inclusion in the study or anamnestic evidence of alcoholism, drug abuse, or medicine abuse.
16. Smoking.
17. Positive blood tests for antibodies to human immunodeficiency virus (HIV) type 1 and 2, antibodies to Treponema pallidum antigens, hepatitis B surface antigen (HBsAg), antibodies to hepatitis C virus antigens, laboratory examination of biomaterial (nasopharyngeal swab) for SARS-Cov-2 RNA (COVID-19).
18. Clinically significant abnormalities on electrocardiogram (ECG).
19. Positive urinalysis for narcotics and powerful drugs.
20. Positive breath alcohol vapor test.
21. Scheduling an inpatient stay during the study period, for any reason other than hospitalization required by this protocol.
22. Failure or inability to comply with protocol requirements, perform protocol-prescribed procedures, diet, and activity regimen.
23. Observance of a religious fast or special diet (e.g., vegetarian, vegan).
24. Other conditions that, in the opinion of the Investigator, preclude a volunteer from enrolling in the study or may result in early withdrawal from the study, including special lifestyles (night work, extreme physical activity).

Withdrawal criteria:

1. The volunteer's refusal to further participate in the study.
2. Failure of the volunteer to comply with the rules of participation in the study (skipping study procedures, independent use of drugs prohibited in the study, violation of dietary and lifestyle restrictions, etc.).
3. Occurrence of causes/occurrence during the study of situations that threaten the safety of the volunteer (e.g., hypersensitivity reactions, etc.).
4. Volunteers included in the study in violation of the inclusion/inclusion criteria.
5. Development of a severe and/or serious adverse event (AE) in a volunteer during the study.
6. Missing 2 or more consecutive blood samples or 3 or more blood samples during one Period of the pharmacokinetic portion of the study.
7. Occurrence of vomiting/diarrhea within 24 h of study drug administration (the choice of time interval is based on the tmax parameter value for doxylamine and pyridoxal-5-phosphate not exceeding 7.2 ± 1.9 and 11.7 ± 5.3 h, respectively, according to the manufacturer of the reference drug).
8. Positive urine test for narcotic substances and potent drugs.
9. Positive breath alcohol vapor test.
10. A positive pregnancy test.
11. Positive test for SARS-Cov-2 RNA (COVID-19);
12. Other causes occurring in the course of the study that prevent the study from being conducted according to the protocol.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - Cmax (Doxylamine) | From 0 to 72 hours (Day 1-4 and Day 22-25)
  Maximum plasma concentration (Cmax)
Pharmacokinetics - Cmax (Pyridoxal-5-phosphate) | From 0 to 72 hours (Day 1-4 and Day 22-25)
  Maximum plasma concentration (Cmax)
Pharmacokinetics - tmax (Doxylamine) | From 0 to 72 hours (Day 1-4 and Day 22-25)
  Time to reach Cmax (tmax)
Pharmacokinetics - tmax (Pyridoxal-5-phosphate) | From 0 to 72 hours (Day 1-4 and Day 22-25)
  Time to reach Cmax (tmax)
Pharmacokinetics - AUC0-t (Doxylamine) | From 0 to 72 hours (Day 1-4 and Day 22-25)
  Area under the plasma concentration-time curve from time 0 to t (AUC0-t)
Pharmacokinetics - AUC0-t (Pyridoxal-5-phosphate) | From 0 to 72 hours (Day 1-4 and Day 22-25)
  Area under the plasma concentration-time curve from time 0 to t (AUC0-t)
Pharmacokinetics - AUC0-inf (Doxylamine) | From 0 to 72 hours (Day 1-4 and Day 22-25)
  Area under the plasma concentration-time curve from time 0 to infinity (AUC0-inf)
Pharmacokinetics - AUC0-inf (Pyridoxal-5-phosphate) | From 0 to 72 hours (Day 1-4 and Day 22-25)
  Area under the plasma concentration-time curve from time 0 to infinity (AUC0-inf)
Pharmacokinetics - AUCextr (Doxylamine) | From 0 to 72 hours (Day 1-4 and Day 22-25)
  Extrapolated AUC, defined as (AUC0-inf - AUC0-t)/AUC0-inf
Pharmacokinetics - AUCextr (Pyridoxal-5-phosphate) | From 0 to 72 hours (Day 1-4 and Day 22-25)
  Extrapolated AUC, defined as (AUC0-inf - AUC0-t)/AUC0-inf
Pharmacokinetics - t1/2 (Doxylamine) | From 0 to 72 hours (Day 1-4 and Day 22-25)
  Elimination half-life (t1/2)
Pharmacokinetics - t1/2 (Pyridoxal-5-phosphate) | From 0 to 72 hours (Day 1-4 and Day 22-25)
  Elimination half-life (t1/2)
Pharmacokinetics - kel (Doxylamine) | From 0 to 72 hours (Day 1-4 and Day 22-25)
  Elimination constant (kel)
Pharmacokinetics - kel (Pyridoxal-5-phosphate) | From 0 to 72 hours (Day 1-4 and Day 22-25)
  Elimination constant (kel)
Pharmacokinetics - MRT (Doxylamine) | From 0 to 72 hours (Day 1-4 and Day 22-25)
  Mean residence time (MRT)
Pharmacokinetics - MRT (Pyridoxal-5-phosphate) | From 0 to 72 hours (Day 1-4 and Day 22-25)
  Mean residence time (MRT)
Bioequivalence - ratio of Cmax (Doxylamine) | From 0 to 72 hours (Day 1-4 and Day 22-25)
  Ratio of geometric mean Cmax after intake of R or T (with 90% confidence intervals)
Bioequivalence - ratio of Cmax (Pyridoxal-5-phosphate) | From 0 to 72 hours (Day 1-4 and Day 22-25)
  Ratio of geometric mean Cmax after intake of R or T (with 90% confidence intervals)
Bioequivalence - ratio of AUC0-t (Doxylamine) | From 0 to 72 hours (Day 1-4 and Day 22-25)
  Ratio of geometric mean AUC0-t after intake of R or T (with 90% confidence intervals)
Bioequivalence - ratio of AUC0-t (Pyridoxal-5-phosphate) | From 0 to 72 hours (Day 1-4 and Day 22-25)
  Ratio of geometric mean AUC0-t after intake of R or T (with 90% confidence intervals)
Bioequivalence - ratio of AUC0-inf (Doxylamine) | From 0 to 72 hours (Day 1-4 and Day 22-25)
  Ratio of geometric mean AUC0-inf after intake of R or T (with 90% confidence intervals)
Bioequivalence - ratio of AUC0-inf (Pyridoxal-5-phosphate) | From 0 to 72 hours (Day 1-4 and Day 22-25)
  Ratio of geometric mean AUC0-inf after intake of R or T (with 90% confidence intervals)

SECONDARY OUTCOMES:
Safety and Tolerability: adverse event (AE) number and frequency | From the screening (and signing informed consent form) to Day 29 of the study or to an early termination visit within the time frame of the study (from Day 0 to Day 29)
  Number and frequency of adverse events (AEs)
serious adverse event (SAE) number and frequency | From the screening (and signing informed consent form) to Day 29 of the study or to an early termination visit within the time frame of the study (from Day 0 to Day 29)
  Number and frequency of serious AEs (SAEs)
Safety and Tolerability: vital signs - systolic blood pressure (SBP) | Screening, from Day 0 to Day 4, from Day 21 to Day 25, and/or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  SBP, mmHg
Safety and Tolerability: vital signs - diastolic blood pressure (DBP) | Screening, from Day 0 to Day 4, from Day 21 to Day 25, and/or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  DBP, mmHg
Safety and Tolerability: vital signs - respiratory rate (RR) | Screening, from Day 0 to Day 4, from Day 21 to Day 25, and/or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  RR, breaths per minute
Safety and Tolerability: vital signs - heart rate (HR) | Screening, from Day 0 to Day 4, from Day 21 to Day 25, and/or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  HR, beats per minute
Safety and Tolerability: vital signs - body temperature | Screening, from Day 0 to Day 4, from Day 21 to Day 25, and/or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Body temperature, centigrade scale
Safety and Tolerability: physical examination results | Screening, from Day 0 to Day 4, from Day 21 to Day 25, and/or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Physical examination will follow the general rules of internal medicine: general examination, examination of mucous membranes and skin, including palpation of lymph nodes, evaluation of the musculoskeletal system, palpation, percussion, and auscultation of the main organ systems (cardiovascular, respiratory, digestive, and urinary systems) will be performed sequentially.
Safety and Tolerability: 12-lead electrocardiogram (ECG) - heart rate | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: heart rate (beats per minute)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - PQ interval | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: PQ interval (ms)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - QRS complex | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: QRS complex (ms)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - corrected QT interval (QTc) | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: QTc (ms)
Safety and Tolerability: urinalysis - color | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Color of the urine
Safety and Tolerability: urinalysis - transparency | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Transparency of the urine
Safety and Tolerability: urinalysis - pH | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  pH of the urine
Safety and Tolerability: urinalysis - specific gravity | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Specific gravity of the urine
Safety and Tolerability: urinalysis - protein | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Protein in the urine (g/L)
Safety and Tolerability: urinalysis - glucose | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Glucose in the urine (mmol/L)
Safety and Tolerability: urinalysis (microscopy) - red blood cells | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Red blood cells in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - white blood cells | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  White blood cells in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - epithelial cells | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Epithelial cells in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - cylinders | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Cylinders in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - mucus | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Mucus in the urine (presence in sight)
Safety and Tolerability: urinalysis (microscopy) - bacteria | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Bacteria in the urine (number in sight)
Safety and Tolerability: complete blood count - hemoglobin | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Hemoglobin, g/dL
Safety and Tolerability: complete blood count - red blood cells | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Red blood cells, 10^6/uL
Safety and Tolerability: complete blood count - hematocrit | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Hematocrit, %
Safety and Tolerability: complete blood count - platelets | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Platelets, 10^3/uL
Safety and Tolerability: complete blood count - white blood cells | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  White blood cells, 10^3/uL
Safety and Tolerability: complete blood count - erythrocyte sedimentation rate | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Erythrocyte sedimentation rate, mm per hour
Safety and Tolerability: complete blood count - neutrophils | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Neutrophils, %
Safety and Tolerability: complete blood count - lymphocytes | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Lymphocytes, %
Safety and Tolerability: complete blood count - eosinophils | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Eosinophils, %
Safety and Tolerability: complete blood count - monocytes | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Monocytes, %
Safety and Tolerability: complete blood count - basophils | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Basophils, %
Safety and Tolerability: blood test results - total protein | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Total protein in blood serum, g/L
Safety and Tolerability: blood test results - creatinine | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Creatinine in blood serum, umol/L
Safety and Tolerability: blood test results - glucose | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Glucose in blood serum, mmol/L
Safety and Tolerability: blood test results - total bilirubin | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Total bilirubin in blood serum, umol/L
Safety and Tolerability: blood test results - total cholesterol | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  Total cholesterol in blood serum, mmol/L
Safety and Tolerability: blood test results - alanine transaminase (ALT) | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  ALT in blood serum, U/L
Safety and Tolerability: blood test results - aspartate transaminase (AST) | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  AST in blood serum, U/L
Safety and Tolerability: blood test results - alkaline phosphatase (ALP) | Screening, Day 4, Day 25 or on early termination visit within the time frame of the study (from Day 0 to Day 29)
  ALP in blood serum, U/L

CONTACTS AND LOCATIONS:
Locations (1):
- Llc "Certa Clinic", Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided